CLINICAL TRIAL: NCT01975324
Title: Dalfampridine Treatment for Nonarteritic Anterior Ischemic Optic Neuropathy (NAION)
Brief Title: A New Medicine to Treat Nonarteritic Anterior Ischemic Optic Neuropathy (NAION)
Acronym: Ampyra
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neuro-Ophthalmologic Associates, PC (Other)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Principal Investigator, Mark L. Moster, M.d., Neuro-Ophthalmologist, Neuro-Ophthalmologic Associates, PC
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Dalfampridine 13-265
Record Dates: First submitted 2013-07-26; First posted 2013-11-04 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-10

CONDITIONS: Non Arteritic Ischemic Optic Neuropathy
Keywords: Ampyra; NAION; Dalfampridine
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — 4-Aminopyridine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dalfampridine (ampyra) (Experimental): Dalfampridine (ampyra) 10mgs twice a day (b.i.d.)for two weeks
  Interventions: Drug: dalfampridine
- Placebo (Placebo Comparator): placebo (sugar Pill) twice a day (b.i.d.)for two weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dalfampridine — dalfampridine 10 mgs or placebo twice a day for two weeks, wash out period of two weeks, dalfampridine 10mgs or placebo twice a day for two weeks
  Other Names: Ampyra
  Arms: dalfampridine (ampyra)
Drug: Placebo — placebo (sugar pill) twice a day for two weeks
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Determine whether dalfampridine (Ampyra) can improve visual function in patients who have had nonarteritic ischemic optic neuropathy (NAION) with stable visual impairment.

DETAILED DESCRIPTION:
The aim of this study is to determine whether dalfampridine can improve visual function in patients who have had nonarteritic ischemic optic neuropathy (NAION) with stable visual impairment.

The objective of this double masked crossover study is to determine whether visual function can be improved in numerous parameters. This includes high contrast visual acuity, low contrast visual acuity, visual field, visual quality of life (VFQ-39), electrophysiology, multi focal electro retinography (mERG), visual evoked potential (VEP), and structure, spectral domain optical coherence tomography (OCT).

Based on the promising results of the use of dalfampridine in Multiple Sclerosis (MS) and in stroke, we hypothesize that the patients with chronic stable deficits after nonarteritic ischemic optic neuropathy (NAION) will have improved visual function with the administration of dalfampridine.

ELIGIBILITY:
Inclusion Criteria:

* NAION 6 months prior to enrollment
* visual acuity of 20/40 or worse

Exclusion Criteria:

Current use of Dalfampridine (Ampyra)

* Pregnancy
* History of seizures
* Renal Failure
* Not able to perform testing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improve visual function | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Moster, MD, Principal Investigator — Neuro-Ophthalmologic Associates, PC
Locations (1):
- Neuro-Ophthalmologic Associates, PC, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newman NJ, Scherer R, Langenberg P, Kelman S, Feldon S, Kaufman D, Dickersin K; Ischemic Optic Neuropathy Decompression Trial Research Group. The fellow eye in NAION: report from the ischemic optic neuropathy decompression trial follow-up study. Am J Ophthalmol. 2002 Sep;134(3):317-28. doi: 10.1016/s0002-9394(02)01639-2. PMID 12208242
- [Background] The ischemic optic neuropathy decompression trial (IONDT): design and methods. Control Clin Trials. 1998 Jun;19(3):276-96. doi: 10.1016/s0197-2456(98)00003-8. PMID 9620811
- [Background] Bever CT Jr. 10 questions about 4-aminopyridine and the treatment of multiple sclerosis. Neurologist. 2009 May;15(3):161-2. doi: 10.1097/NRL.0b013e3181679be5. No abstract available. PMID 19430274
- [Background] Davis FA, Stefoski D, Rush J. Orally administered 4-aminopyridine improves clinical signs in multiple sclerosis. Ann Neurol. 1990 Feb;27(2):186-92. doi: 10.1002/ana.410270215. PMID 2317014
- [Background] Jones RE, Heron JR, Foster DH, Snelgar RS, Mason RJ. Effects of 4-aminopyridine in patients with multiple sclerosis. J Neurol Sci. 1983 Aug-Sep;60(3):353-62. doi: 10.1016/0022-510x(83)90145-4. PMID 6631441
- [Background] Stefoski D, Davis FA, Faut M, Schauf CL. 4-Aminopyridine improves clinical signs in multiple sclerosis. Ann Neurol. 1987 Jan;21(1):71-7. doi: 10.1002/ana.410210113. PMID 2435223
- [Background] van Diemen HA, van Dongen MM, Dammers JW, Polman CH. Increased visual impairment after exercise (Uhthoff's phenomenon) in multiple sclerosis: therapeutic possibilities. Eur Neurol. 1992;32(4):231-4. doi: 10.1159/000116830. PMID 1324180
- [Background] Bever CT Jr, Young D, Anderson PA, Krumholz A, Conway K, Leslie J, Eddington N, Plaisance KI, Panitch HS, Dhib-Jalbut S, et al. The effects of 4-aminopyridine in multiple sclerosis patients: results of a randomized, placebo-controlled, double-blind, concentration-controlled, crossover trial. Neurology. 1994 Jun;44(6):1054-9. doi: 10.1212/wnl.44.6.1054. PMID 8208399
- [Background] Stefoski D, Davis FA, Fitzsimmons WE, Luskin SS, Rush J, Parkhurst GW. 4-Aminopyridine in multiple sclerosis: prolonged administration. Neurology. 1991 Sep;41(9):1344-8. doi: 10.1212/wnl.41.9.1344. PMID 1891078
- [Background] Polman CH, Bertelsmann FW, de Waal R, van Diemen HA, Uitdehaag BM, van Loenen AC, Koetsier JC. 4-Aminopyridine is superior to 3,4-diaminopyridine in the treatment of patients with multiple sclerosis. Arch Neurol. 1994 Nov;51(11):1136-9. doi: 10.1001/archneur.1994.00540230074016. PMID 7980110
- [Background] Strupp M, Brandt T. Pharmacological advances in the treatment of neuro-otological and eye movement disorders. Curr Opin Neurol. 2006 Feb;19(1):33-40. doi: 10.1097/01.wco.0000196156.00481.e1. PMID 16415675
- [Background] Goodman AD, Brown TR, Krupp LB, Schapiro RT, Schwid SR, Cohen R, Marinucci LN, Blight AR; Fampridine MS-F203 Investigators. Sustained-release oral fampridine in multiple sclerosis: a randomised, double-blind, controlled trial. Lancet. 2009 Feb 28;373(9665):732-8. doi: 10.1016/S0140-6736(09)60442-6. PMID 19249634
- [Background] Goodman AD, Brown TR, Edwards KR, Krupp LB, Schapiro RT, Cohen R, Marinucci LN, Blight AR; MSF204 Investigators. A phase 3 trial of extended release oral dalfampridine in multiple sclerosis. Ann Neurol. 2010 Oct;68(4):494-502. doi: 10.1002/ana.22240. PMID 20976768
- [Background] Ho PW, Reutens DC, Phan TG, Wright PM, Markus R, Indra I, Young D, Donnan GA. Is white matter involved in patients entered into typical trials of neuroprotection? Stroke. 2005 Dec;36(12):2742-4. doi: 10.1161/01.STR.0000189748.52500.a7. Epub 2005 Nov 3. PMID 16269640